CLINICAL TRIAL: NCT05186584
Title: Effects of Maitland's Antero-posterior Versus Lateral Mobilizations on Cardiovascular Responses in Non-Specific Chronic Neck Pain
Brief Title: Effects of Maitland's Antero-Posterior Versus Lateral Mobilizations on Cardiovascular Responses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ayesha Afsar
Record Dates: First submitted 2021-12-29; First posted 2022-01-11 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Neck Pain
Keywords: Maitland mobilization
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAITLAND'S ANTEROPOSTERIOR(AP) MOBILIZATION (Experimental): Patients in this group will receive Maitland's Antero-Posterior Mobilization.
  Interventions: Other: MAITLAND'S ANTEROPOSTERIOR(AP) MOBILIZATION
- MAITLAND'S LATERAL MOBILIZATION (Experimental): Patients in this group will receive Maitland's Lateral Mobilization.
  Interventions: Other: MAITLAND'S LATERAL MOBILIZATION

INTERVENTIONS:
Other: MAITLAND'S ANTEROPOSTERIOR(AP) MOBILIZATION — Group A will receive the 5 sets of 10 seconds Grade 1 mobilizations with a rate of 15 oscillations each set (total 75 oscillations) for AP mobilizations at most symptomatic segment, with 10 seconds rest between sets. Most symptomatic segment is that segment of cervical spine at which patient will feel greatest pain by palpation.
  For AP mobilizations, patient will lye supine and therapist will stand by his head. Therapist will make broad contact with the thumb, at the costal process of the vertebrae to be mobilized and spread fingers around adjacent neck for stability. Shoulder will be positioned above the joint being treated. Gentle oscillatory Anteroposterior pressure will be performed by the therapist's arm and trunk.
  Arms: MAITLAND'S ANTEROPOSTERIOR(AP) MOBILIZATION
Other: MAITLAND'S LATERAL MOBILIZATION — Group B will receive the same sets (i.e. 5 sets of 10 seconds Grade 1 mobilizations with a rate of 15 oscillations each set) for lateral mobilizations at most symptomatic segment, with 10 sec rest between each set. For lateral mobilization, patient will lye supine and therapist will stand by his head. Therapist will place the anterolateral aspect 2nd metacarpophalangeal joint over the lateral aspect of transverse process of most symptomatic segment. Gentle lateral oscillations towards the asymptomatic side will be provided by the therapist.
  Arms: MAITLAND'S LATERAL MOBILIZATION

SUMMARY:
This study will be a randomized control trial and will be conducted in Polyclinic Hospital Islamabad & Rawal Dental and General Hospital Rawalpindi. A sample of 62 participants will be taken. Patients will be divided into two equal groups of 31 participants in each group, group Randomization will be done through flip coin method. Patients in group A will receive Maitland's antero-posterior Mobilization, while Patients in group B will receive Maitland's lateral mobilizations. 4 sessions of treatment will be given for 2 weeks with interval of 3 days, 4 days and 7 days between 1st & 2nd session, 2nd & 3rd session and 3rd & 4th session, respectively. The outcome measures will be OMRON Automatic Blood Pressure Monitor, Numeric pain rating scale(NPRS) and Global Rating of Change questionare will be measured at baseline and at the end of 4th session. Data will be analyzed by SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Age 25 to 55 years
* Pain in neck with no known cause for > 3 months
* Resting systolic blood pressure between 90 to 139 mmHg
* resting diastolic blood pressure between 60 to 88 mmHg
* resting heart rate between 60 to 100 beats/min
* no prior exposure to antero-posterior and lateral mobilizations

Exclusion Criteria:

* Participants falling in this category would be excluded from the study.
* age <25 and >55
* current smokers
* history of fainting spells, diabetes mellitus, spinal surgery and whiplash injury( in last 6 months)
* taking medications for blood thinning, diabetes mellitus
* having neurologic or cardiovascular disease, radiating pain, cervicogenic headaches
* movement coordination impairment
* athletes
* unable to read and write

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
OMRON Automatic Blood Pressure Monitor | 2 Weeks
  The Omron is an automatic digital device for professional blood pressure measurement at the upper arm level. It measures BP range of 0-299 mmHg
OMRON Automatic heart rate Monitor | 2 Weeks
  The Omron is an automatic digital device for professional heart rate range of 40 -180 beats/min
Numeric Pain Rating Scale (NPRS) | 2 Weeks
  It is a tool used for measuring intensity of pain. Patient select numeric from (0-10) that reflects his/her pain intensity. The reliability of tool is ICC = 0.67; [0.27 to 0.84])
Global Rating of Change (GROC) | 2 Weeks
  It is a scale commonly used in clinical research, particularly in the musculoskseletal area to measure a patient's improvement or deterioration over time, to determine the eﬀect of an intervention .

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Rawal General Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No